CLINICAL TRIAL: NCT00175877
Title: A Phase III Multi-centre, Open-label, follow-on Study to CDP870-027, to Assess the Efficacy and Safety of Lyophilized CDP870 an Engineered Human Anti-TNF PEG Conjugate, as Additional Medication to Methotrexate, in the Treatment of Signs and Symptoms and Preventing Structural Damage in Patients With Active Rheumatoid Arthritis
Brief Title: A Study of the Safety and Effectiveness of Lyophilized Certolizumab Pegol in the Treatment of Signs and Symptoms of Rheumatoid Arthritis and in Prevention of Joint Damage in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87028; 2005-001350-24 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; CDP870; Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab Pegol (Experimental): All patients received Certolizumab Pegol (CZP) 400 mg subcutaneously (sc) every two weeks, given as two 1 ml injections of CZP for at least six months and then 200 mg of CZP sc every two weeks, given as one 1 ml injection.
  Interventions: Biological: Certolizumab Pegol

INTERVENTIONS:
Biological: Certolizumab Pegol — Strength and Form: Lyophilized product reconstituted to 1 ml containing 200 mg of Certolizumab Pegol (CZP) given as a subcutaneous injection.
  Dosage and Frequency: 400 mg every two weeks for at least 6 months, then 200 mg every two weeks.
  Duration: Until end of study.
  Other Names: Cimzia

SUMMARY:
An open ended study in which patients who completed the double-blind study CDP870-027 [NCT00152386] are given Certolizumab Pegol (CZP) and assessed for signs and symptoms of Rheumatoid Arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

Patients must have either failed to achieve American College of Rheumatology 20 % Response Criteria (ACR20) at Weeks 12 and 14 in C87027 [NCT00152386], or must have completed the entire Week 52 assessment of C87027 [NCT00152386] trial.

Exclusion Criteria:

* A diagnosis of any other inflammatory Arthritis (e.g. Psoriatic Arthritis or Ankylosing Spondylitis)
* A secondary, non-inflammatory type of Arthritis (e.g. Osteoarthritis or Fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with evaluation of the effect of CDP870 on the patient's primary diagnosis of Rheumatoid Arthritis
* Any concomitant biological therapy
* Any experimental therapy, within or outside a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 857 (Actual)
Dates: Start 2005-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (121):
- United States (19):
  - 152, Huntsville, Alabama
  - 148, San Diego, California
  - 153, Danbury, Connecticut
  - 133, Ocala, Florida
  - 140, Orlando, Florida
  - 150, Orlando, Florida
  - 145, Sarasota, Florida
  - 136, Tampa, Florida
  - 157, Coeur d'Alene, Idaho
  - 155, Springfield, Illinois
  - 134, Wheaton, Maryland
  - 151, St Louis, Missouri
  - 156, Lincoln, Nebraska
  - 135, Charlotte, North Carolina
  - 147, Cleveland, Ohio
  - 158, Dayton, Ohio
  - 139, Charleston, South Carolina
  - 137, Austin, Texas
  - 143, San Antonio, Texas
- Argentina (11):
  - 12, Buenos Aires
  - 14, Capital Federal
  - 1, Capital Federal
  - 9, Capital Federal
  - 8, Ciudad Autonoma de Buenos Aire
  - 11, Córdoba
  - 2, Córdoba
  - 13, Quilmes
  - 7, Rosario
  - 10, San Miguel de Tucumán
  - 6, Santa Fe
- Australia (3):
  - 18, Malvern
  - 21, Maroochydore
  - 23, Perth
- Belgium (3):
  - 179, Antwerp
  - 199, Liège
  - 177, Merksem
- Bulgaria (5):
  - 29, Pleven
  - 221, Sofia
  - 28, Sofia
  - 30, Sofia
  - 26, Stara Zagora
- Canada (8):
  - 43, Newmarket, Ontario
  - 32, Toronto, Ontario
  - 39, Toronto, Ontario
  - 35, Hamilton
  - 36, Kitchener
  - 201, Pointe-Claire
  - 31, Sainte-Foy
  - 203, Winnipeg
- Chile (3):
  - 190, Santiago
  - 49, Santiago
  - 44, Valdivia
- 52, Rijeka, Croatia
- Czechia (8):
  - 56, Brno
  - 57, Ostrava Trebovice
  - 187, Pilsen
  - 55, Prague
  - 60, Prague
  - 61, Prague
  - 58, Uherské Hradiště
  - 62, Zlín
- Estonia (3):
  - 64, Pärnu
  - 65, Tallinn
  - 63, Tartu
- 68, Hyvinkää, Finland
- 160, Montpellier, France
- Hungary (6):
  - 71, Budapest
  - 73, Budapest
  - 75, Bupadest
  - 191, Debrecen
  - 76, Miskolc
  - 74, Szolnok
- Israel (7):
  - 79, Afula
  - 82, Ashkelon
  - 81, Haifa
  - 83, Haifa
  - 78, Ramat Gan
  - 77, Tel Aviv
  - 85, Ẕerifin
- Latvia (2):
  - 86, Riga
  - 88, Riga
- Lithuania (6):
  - 92, Alytus
  - 89, Kaunas
  - 91, Klaipėda
  - 93, Panevezys
  - 90, Šiauliai
  - 94, Vilnius
- Mexico (2):
  - 95, Mexicalli
  - 96, Monterrey
- New Zealand (4):
  - 103, Auckland
  - 101, Christchurch
  - 100, South Canterbury
  - 192, Tauranga
- Russia (10):
  - 107, Moscow
  - 113, Moscow
  - 222, Moscow
  - 223, Moscow
  - 224, Moscow
  - 109, Saint Petersburg
  - 111, Saint Petersburg
  - 112, Saint Petersburg
  - 193, Saint Petersburg
  - 110, Yaroslavl
- Serbia (4):
  - 117, Belgrade
  - 118, Belgrade
  - 114, Niška Banja
  - 115, Novi Sad
- Slovakia (4):
  - 119, Bratislava
  - 121, Košice
  - 120, Piešťany
  - 122, Piešťany
- Ukraine (10):
  - 210, Dnipro
  - 209, Donetsk
  - 216, Donetsk
  - 213, Ivano-Frankivsk
  - 211, Kiev
  - 212, Kiev
  - 215, Kiev
  - 220, Kiev
  - 208, Symferopyl
  - 214, Zaporizhzhya

REFERENCES:
- [Background] Paul S, Marotte H, Kavanaugh A, Goupille P, Kvien TK, de Longueville M, Mulleman D, Sandborn WJ, Vande Casteele N. Exposure-Response Relationship of Certolizumab Pegol and Achievement of Low Disease Activity and Remission in Patients With Rheumatoid Arthritis. Clin Transl Sci. 2020 Jul;13(4):743-751. doi: 10.1111/cts.12760. Epub 2020 Apr 1. PMID 32100960
- [Result] Keystone EC, Combe B, Smolen J, Strand V, Goel N, van Vollenhoven R, Mease P, Landewe R, Fleischmann R, Luijtens K, van der Heijde D. Sustained efficacy of certolizumab pegol added to methotrexate in the treatment of rheumatoid arthritis: 2-year results from the RAPID 1 trial. Rheumatology (Oxford). 2012 Sep;51(9):1628-38. doi: 10.1093/rheumatology/kes082. Epub 2012 May 16. PMID 22596211
- [Result] van der Heijde D, Keystone EC, Curtis JR, Landewe RB, Schiff MH, Khanna D, Kvien TK, Ionescu L, Gervitz LM, Davies OR, Luijtens K, Furst DE. Timing and magnitude of initial change in disease activity score 28 predicts the likelihood of achieving low disease activity at 1 year in rheumatoid arthritis patients treated with certolizumab pegol: a post-hoc analysis of the RAPID 1 trial. J Rheumatol. 2012 Jul;39(7):1326-33. doi: 10.3899/jrheum.111171. Epub 2012 May 15. PMID 22589265
- [Result] Curtis JR, Chen L, Luijtens K, Navarro-Millan I, Goel N, Gervitz L, Weinblatt M. Dose escalation of certolizumab pegol from 200 mg to 400 mg every other week provides no additional efficacy in rheumatoid arthritis: an analysis of individual patient-level data. Arthritis Rheum. 2011 Aug;63(8):2203-8. doi: 10.1002/art.30387. PMID 21484766
- [Derived] Curtis JR, Winthrop K, O'Brien C, Ndlovu MN, de Longueville M, Haraoui B. Use of a baseline risk score to identify the risk of serious infectious events in patients with rheumatoid arthritis during certolizumab pegol treatment. Arthritis Res Ther. 2017 Dec 15;19(1):276. doi: 10.1186/s13075-017-1466-y. PMID 29246162
- [Derived] Smolen J, Landewe RB, Mease P, Brzezicki J, Mason D, Luijtens K, van Vollenhoven RF, Kavanaugh A, Schiff M, Burmester GR, Strand V, Vencovsky J, van der Heijde D. Efficacy and safety of certolizumab pegol plus methotrexate in active rheumatoid arthritis: the RAPID 2 study. A randomised controlled trial. Ann Rheum Dis. 2009 Jun;68(6):797-804. doi: 10.1136/ard.2008.101659. Epub 2008 Nov 17. PMID 19015207
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of subjects started in June 2005. 121 centers in 22 countries enrolled subjects.
  Participant Flow refers to the Safety Set consisting of all enrolled subjects who received at least 1 dose of study medication.
  Of the 857 enrolled subjects, 846 subjects are included in the Safety Set. There was 1 enrolled subject who was never dosed.
Pre-assignment Details: The study consists of 2 populations: of subjects who failed to achieve predefined criteria in preceding study NCT00152386 who entered C87028 on Week 16 of preceding study and of those who completed Week 52 of preceding study.
  Due to findings of fraud at one site, data of the 10 subjects of the site were not analyzed with data from other sites.
Groups:
- Certolizumab Pegol: All patients received Certolizumab Pegol (CZP) 400 mg subcutaneously (sc) every two weeks, given as two 1 ml injections of CZP for at least six months and then 200 mg of CZP sc every two weeks, given as one 1 ml injection.
  Certolizumab Pegol : Strength and Form: Lyophilized product reconstituted to 1 ml containing 200 mg of Certolizumab Pegol (CZP) given as a subcutaneous injection.
  Dosage and Frequency: 400 mg every two weeks for at least 6 months, then 200 mg every two weeks.
  Duration: Until end of study.
Period: Overall Study
Arm/Group | Certolizumab Pegol
Started | 846
Completed | 497
Not Completed | 349
Not completed — Adverse Event | 136
Not completed — Withdrawal by Subject | 141
Not completed — Lost to Follow-up | 9
Not completed — Lack of Efficacy | 26
Not completed — Protocol Violation | 15
Not completed — Other Reason | 20
Not completed — AE & Other | 1
Not completed — Withdrawal by subject & Other | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS). SS consists of all enrolled subjects who received at least 1 dose of study medication.
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 846
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 736
  >=65 years | 109
Age, Continuous [Mean (Full Range); unit: years] | 51.5 (11.4) [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 701
  Male | 145
Region of Enrollment [Number; unit: participants]
  Serbia | 45
  United States | 56
  Estonia | 16
  Slovakia | 45
  Finland | 5
  Ukraine | 81
  Lithuania | 42
  Russian Federation | 102
  Israel | 24
  Chile | 11
  France | 2
  Czech Republic | 122
  Hungary | 57
  Mexico | 5
  Canada | 19
  Argentina | 122
  Belgium | 5
  Croatia | 3
  Australia | 12
  Bulgaria | 28
  Latvia | 26
  New Zealand | 18
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 73.69 (16.17)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 164.30 (8.88)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Adverse Event (AE) From First Certolizumab Pegol (CZP) Dose up to Approximately 7 Years
Description: An AE is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
  First dose of Certolizumab Pegol (CZP) was at Baseline of the preceding double-blind study [NCT00152386] for subjects randomized to CZP, or at Entry Visit (Week 0) of this study for subjects randomized to Placebo.
Time Frame: From first dose of CZP to the end of the open-label study (approximately 7 years)
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 846
percentage of participants | 94.9

2. Primary Outcome: Percentage of Subjects With at Least One Serious Adverse Event (SAE) From First Certolizumab Pegol (CZP) Dose up to Approximately 7 Years
Description: A SAE is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly or birth defect
  * Is as infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardise the patients, or may require medical or surgical intervention to prevent any of the above
  First dose of CZP was at Baseline of the preceding double-blind study [NCT00152386] for subjects randomized to CZP, or at Entry Visit (Week 0) of this study for subjects randomized to Placebo.
Time Frame: From first dose of CZP to the end of the open-label study (approximately 7 years)
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 846
percentage of participants | 41.6

3. Primary Outcome: Percentage of Subjects Who Withdrew Due to an Adverse Event (AE) During the Study
Description: An AE is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage. The results of this Primary Outcome Measure are summarized from the Adverse Event pages of the Case Report Forms.
Time Frame: From Entry Visit (Week 0) to the end of the study (approximately 6.5 years)
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 846
percentage of participants | 16.2

4. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 48
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 48 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 48 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 733 are included in this analysis. Data not available for 113 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 733
percentage of participants | 87.0 [84.4 to 89.4]

5. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 96
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 96 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 96 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 668 are included in this analysis. Data not available for 178 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 668
percentage of participants | 88.0 [85.3 to 90.4]

6. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 144
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 144 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 144 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 602 are included in this analysis. Data not available for 244 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 602
percentage of participants | 87.9 [85.0 to 90.4]

7. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 192
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 192 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 192 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 537 are included in this analysis. Data not available for 309 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 537
percentage of participants | 89.4 [86.5 to 91.9]

8. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 240
Description: The assessments are based on a 20 % or greater improvement from Baseline to Week 240 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 240 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 183 are included in this analysis. Data not available for 663 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 183
percentage of participants | 82.5 [76.2 to 87.7]

9. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Completion/Withdrawal
Description: The assessments are based on a 20 % or greater improvement from Baseline to Completion/Withdrawal in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Completion/Withdrawal of the open-label study (up to approximately 7 years)
Population: Of the 846 subjects in the Safety Set (SS), 841 are included in this analysis. Data not available for 5 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 841
percentage of participants | 81.3 [78.5 to 83.9]

10. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 48
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 48 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 48 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 733 are included in this analysis. Data not available for 113 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 733
percentage of participants | 63.0 [59.4 to 66.5]

11. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 96
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 96 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 96 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 668 are included in this analysis. Data not available for 178 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 668
percentage of participants | 66.0 [62.3 to 69.6]

12. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 144
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 144 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 144 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 602 are included in this analysis. Data not available for 244 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 602
percentage of participants | 65.4 [61.5 to 69.2]

13. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 192
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 192 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 192 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 537 are included in this analysis. Data not available for 309 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 537
percentage of participants | 64.8 [60.6 to 68.8]

14. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 240
Description: The assessments are based on a 50 % or greater improvement from Baseline to Week 240 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 240 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 183 are included in this analysis. Data not available for 663 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 183
percentage of participants | 58.5 [51.0 to 65.7]

15. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Completion/Withdrawal
Description: The assessments are based on a 50 % or greater improvement from Baseline to Completion/Withdrawal in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: as for outcome 9
Population: Of the 846 subjects in the Safety Set (SS), 841 are included in this analysis. Data not available for 5 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 841
percentage of participants | 57.6 [54.1 to 60.9]

16. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 48
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 48 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 48 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 733 are included in this analysis. Data not available for 113 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 733
percentage of participants | 37.7 [34.1 to 41.3]

17. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 96
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 96 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 96 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 668 are included in this analysis. Data not available for 178 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 668
percentage of participants | 40.7 [37.0 to 44.6]

18. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 144
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 144 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 144 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 602 are included in this analysis. Data not available for 244 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 602
percentage of participants | 41.2 [37.2 to 45.2]

19. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 192
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 192 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 192 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 537 are included in this analysis. Data not available for 309 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 537
percentage of participants | 42.8 [38.6 to 47.1]

20. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 240
Description: The assessments are based on a 70 % or greater improvement from Baseline to Week 240 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: From Baseline of the preceding double-blind study to Week 240 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 183 are included in this analysis. Data not available for 663 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 183
percentage of participants | 34.4 [27.6 to 41.8]

21. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Completion/Withdrawal
Description: The assessments are based on a 70 % or greater improvement from Baseline to Completion/Withdrawal in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP). Baseline is Baseline of the preceding double-blind study.
Time Frame: as for outcome 9
Population: Of the 846 subjects in the Safety Set (SS), 841 are included in this analysis. Data not available for 5 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 841
percentage of participants | 38.2 [34.9 to 41.5]

22. Secondary Outcome: Change From Baseline of the Preceding Double-Blind Study to Week 96 in Modified Total Sharp Score (mTSS)
Description: The mTSS quantifies the extent of bone erosions and joint space narrowing for 44 and 42 joints, respectively, as assessed by x-rays of the hands and feet. The score ranges from 0 to 448 with higher scores representing greater damage. A negative value in mTSS change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: From Baseline of the preceding double-blind study to Week 96 of the open-label study
Population: Of the 846 subjects in the Safety Set (SS), 661 are included in this analysis. Data not available for 185 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 661
units on a scale | 0.95 (4.79)

23. Secondary Outcome: Change From Baseline of the Preceding Double-Blind Study to Completion/Withdrawal Visit in Health Assessment Questionnaire - Disability Index (HAQ-DI) Total Score
Description: The HAQ-DI assesses the degree of difficulty experienced in eight domains (Dressing and Grooming, Arising, Eating, Walking, Hygiene, Reach, Gripping, Other Activities) of daily living activities using 20 questions. The HAQ-DI is calculated by summing the domain scores and dividing them by the number of domains. It ranges from 0 (no difficulty) to 3 (unable to do). Negative values indicate an improvement from Baseline to the Post-Baseline Visit with larger negative values showing a better improvement.
Time Frame: as for outcome 9
Population: Of the 846 subjects in the Safety Set (SS), 824 are included in this analysis. Data not available for 22 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 824
units on a scale | -0.674 (0.640)

24. Secondary Outcome: Change From Baseline to Completion/Withdrawal Visit in Duration of Morning Stiffness
Description: Morning stiffness is defined as the time in hours elapsed between the time of usual awakening (even if not in the morning) and the time the subject is as limber as he/she will be during a day involving typical activities. A negative value in duration of morning stiffness change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: as for outcome 9
Population: Of the 846 subjects in the Safety Set (SS), 838 are included in this analysis. Data not available for 8 subjects.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 838
hours | -2.147 (3.846)

25. Secondary Outcome: Change From Baseline to Completion/Withdrawal Visit in Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28[ESR])
Description: DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. A negative value in DAS28[ESR] change from Baseline indicates an improvement from Baseline.
Time Frame: as for outcome 9
Population: Of the 846 subjects in the Safety Set (SS), 834 are included in this analysis. Data not available for 12 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 834
units on a scale | -3.222 (1.511)

26. Secondary Outcome: Percentage of Subjects With Good European League Against Rheumatism (EULAR) Response at Completion/Withdrawal Visit
Description: Good EULAR response is defined as Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28[ESR]) improvement from Baseline of the preceding double-blind study > 1.2 and DAS28[ESR] value < 3.2.
Time Frame: as for outcome 9
Population: Of the 846 subjects in the Safety Set (SS), 834 are included in this analysis. Data not available for 12 subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 834
percentage of participants | 42.4

27. Secondary Outcome: Change From Baseline to Completion/Withdrawal Visit in Short-Form Health Survey (SF-36) Item Questionnaire Physical Component Summary (PCS) Score
Description: The SF-36 is a 36-item generic health status measure that measures 8 general health concepts: Physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each domain of the eight domains and the summary concept PCS score are scored to yield values between 0 (worst) and 100 (best).
Time Frame: as for outcome 9
Population: Of the 846 subjects in the Safety Set (SS), 777 are included in this analysis. Data not available for 69 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 777
units on a scale | 8.813 (9.092)

28. Secondary Outcome: Change From Baseline to Completion/Withdrawal Visit in Short-Form Health Survey (SF-36) Item Questionnaire Mental Component Summary (MCS) Score
Description: The SF-36 is a 36-item generic health status measure that measures 8 general health concepts: Physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each domain of the eight domains and the summary concept MCS score are scored to yield values between 0 (worst) and 100 (best).
Time Frame: as for outcome 9
Population: Of the 846 subjects in the Safety Set (SS), 777 are included in this analysis. Data not available for 69 subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 777
units on a scale | 4.612 (12.592)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to approximately 7 years, from first dose of Certolizumab Pegol (CZP) to the end of the open-label study.
Description: AEs refer to the Safety Set. Safety Set includes all enrolled subjects who received at least 1 dose of study medication.
Arm/Group | Certolizumab Pegol
Serious Adverse Events (participants affected / at risk) | 352/846
Other Adverse Events (participants affected / at risk) | 682/846
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=846)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 4 (4)
Angina unstable (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 5 (7)
Myocardial ischaemia (Cardiac disorders) | 3 (3)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrioventricular extrasystoles (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (7)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 4 (5)
Macular hole (Eye disorders) | 1 (2)
Retinal detachment (Eye disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Femoral hernia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (2)
Inguinal hernia (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Megacolon (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Sudden death (General disorders) | 2 (2)
Pyrexia (General disorders) | 5 (5)
Chest pain (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 10 (10)
Hepatic cyst (Hepatobiliary disorders) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 3 (3)
Allergy to arthropod bite (Immune system disorders) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Peritoneal infection (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 6 (6)
Asymptomatic bacteriuria (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 11 (12)
Folliculitis (Infections and infestations) | 1 (1)
Arthritis infective (Infections and infestations) | 2 (2)
Bursitis infective (Infections and infestations) | 3 (3)
Sialoadenitis (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 2 (2)
Otitis media acute (Infections and infestations) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1)
Dacryocystitis infective (Infections and infestations) | 1 (1)
Salpingitis (Infections and infestations) | 1 (1)
Geotrichum infection (Infections and infestations) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 5 (5)
Herpes zoster disseminated (Infections and infestations) | 1 (1)
Histoplasmosis (Infections and infestations) | 1 (1)
Abscess soft tissue (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 3 (3)
Groin abscess (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3)
Wound infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4)
Bronchitis acute (Infections and infestations) | 5 (6)
Bronchitis chronic (Infections and infestations) | 1 (2)
Bronchopneumonia (Infections and infestations) | 2 (2)
Lobar pneumonia (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Obstructive chronic bronchitis with acute exacerbation (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 29 (31)
Pyothorax (Infections and infestations) | 2 (2)
Nocardiosis (Infections and infestations) | 1 (1)
Condyloma acuminatum (Infections and infestations) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 4 (4)
Urosepsis (Infections and infestations) | 2 (2)
Burn infection (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 2 (2)
Pyoderma (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 5 (5)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 6 (6)
Meningitis streptococcal (Infections and infestations) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 4 (4)
Pulmonary tuberculosis (Infections and infestations) | 9 (9)
Tuberculosis (Infections and infestations) | 3 (3)
Tuberculous pleurisy (Infections and infestations) | 2 (2)
Acute sinusitis (Infections and infestations) | 2 (2)
Acute tonsillitis (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (2)
Chronic tonsillitis (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Laryngopharyngitis (Infections and infestations) | 1 (1)
Nasal vestibulitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3)
Tonsillitis (Infections and infestations) | 4 (5)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 4 (5)
Urinary tract infection (Infections and infestations) | 5 (5)
Viral infection (Infections and infestations) | 1 (1)
Yersinia bacteraemia (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 4 (5)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Haemothorax (Injury, poisoning and procedural complications) | 1 (1)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 (1)
Complication of device removal (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (4)
Lower limb fracture (Injury, poisoning and procedural complications) | 6 (6)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Polytraumatism (Injury, poisoning and procedural complications) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 1 (1)
Vertebral injury (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 3 (3)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 5 (5)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Smear cervix abnormal (Investigations) | 1 (1)
Chest X-ray abnormal (Investigations) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (5)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 7 (8)
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower limb deformity (Musculoskeletal and connective tissue disorders) | 1 (3)
Toe deformity (Musculoskeletal and connective tissue disorders) | 3 (3)
Upper limb deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Wrist deformity (Musculoskeletal and connective tissue disorders) | 1 (2)
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint destruction (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (9)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 34 (38)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lip and/ or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vaginal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (5)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (4)
Conversion disorder (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Stress incontinence (Renal and urinary disorders) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 4 (4)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 4 (4)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Ovarian haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 2 (2)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 2 (2)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Alveolitis fibrosing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 3 (3)
Knee arthroplasty (Surgical and medical procedures) | 3 (3)
Synovectomy (Surgical and medical procedures) | 1 (1)
Brain operation (Surgical and medical procedures) | 1 (1)
Therapy regimen changed (Surgical and medical procedures) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 3 (3)
Arteriosclerosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 6 (6)
Trombophlebitis (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 3 (4)
Essential hypertension (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Rheumatoid vasculitis (Vascular disorders) | 2 (2)
Vasculitis (Vascular disorders) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=846)
Anaemia (Blood and lymphatic system disorders) | 57 (77)
Conjunctivitis (Eye disorders) | 55 (77)
Diarrhoea (Gastrointestinal disorders) | 66 (90)
Nausea (Gastrointestinal disorders) | 53 (84)
Dyspepsia (Gastrointestinal disorders) | 57 (76)
Gastritis (Gastrointestinal disorders) | 48 (59)
Pyrexia (General disorders) | 59 (86)
Urinary tract infection (Infections and infestations) | 150 (280)
Nasopharyngitis (Infections and infestations) | 158 (270)
Upper respiratory tract infection (Infections and infestations) | 138 (267)
Bronchitis acute (Infections and infestations) | 99 (134)
Pharyngitis (Infections and infestations) | 86 (132)
Herpes simplex (Infections and infestations) | 71 (131)
Influenza (Infections and infestations) | 87 (115)
Sinusitis (Infections and infestations) | 72 (110)
Bronchitis (Infections and infestations) | 66 (89)
Rhinitis (Infections and infestations) | 56 (75)
Respiratory tract infection (Infections and infestations) | 45 (74)
Hepatic enzyme increased (Investigations) | 45 (73)
Alanine aminotransferase increased (Investigations) | 52 (72)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 133 (225)
Back pain (Musculoskeletal and connective tissue disorders) | 103 (150)
Arthralgia (Musculoskeletal and connective tissue disorders) | 71 (119)
Headache (Nervous system disorders) | 92 (140)
Depression (Psychiatric disorders) | 43 (54)
Cough (Respiratory, thoracic and mediastinal disorders) | 58 (77)
Rash (Skin and subcutaneous tissue disorders) | 63 (84)
Hypertension (Vascular disorders) | 159 (242)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days